CLINICAL TRIAL: NCT03122691
Title: Differences in Cannabis Impairment and Its Measurement Due to Route of Administration
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: RTI International (Other); U.S. Department of Justice (U.S. Federal Agency); National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: IRB00122849; 2016-DN-BX-0193 (Other Grant/Funding Number: National Institute of Justice); R44DA046272-01A1 (NIH); T32DA007209 (NIH)
Record Dates: First submitted 2017-04-17; First posted 2017-04-21 (Actual); Results first posted 2023-02-21 (Actual); Last update posted 2023-02-21 (Actual); Status verified 2023-01

CONDITIONS: Behavioral Pharmacology of Cannabis
MeSH Terms: interventions — nabiximols

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Placebo controlled, double blind drug administration
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Placebo Oral Cannabis (Placebo Comparator): Single acute administration of placebo cannabis baked into a brownie
  Interventions: Drug: cannabis
- Low-Dose Oral Cannabis (Experimental): Single acute administration of cannabis containing 10mg THC baked into a brownie
  Interventions: Drug: cannabis
- High-Dose Oral Cannabis (Experimental): Single acute administration of cannabis containing 25mg THC baked into a brownie
  Interventions: Drug: cannabis
- Placebo Vaporized Cannabis (Placebo Comparator): Single acute administration of placebo cannabis via commercial vaporizer
  Interventions: Drug: cannabis
- Low-Dose Vaporized Cannabis (Experimental): Single acute administration of placebo cannabis containing 5mg THC via commercial vaporizer
  Interventions: Drug: cannabis
- High-Dose Vaporized Cannabis (Experimental): Single acute administration of placebo cannabis containing 20mg THC via commercial vaporizer
  Interventions: Drug: cannabis

INTERVENTIONS:
Drug: cannabis — Cannabis will be self-administered by study participants
  Other Names: marijuana

SUMMARY:
This research is being done to measure the effects of both oral and vaporized cannabis (marijuana), at different doses, on the ability to perform certain tasks such as balancing, eye tracking, and computerized measures of memory and attention, as well as performance on a novel app (DRUID) that is being developed for field sobriety testing. The investigators will collect biological fluids (urine, blood, saliva/spit) after cannabis is eaten or vaporized to see if there are markers in those fluids that can predict performance on the behavioral tasks and the DRUID App. The results of this study will help us better understand the effects of using cannabis, and to help identify behaviors and/or substances in the body that relate to cannabis impairment.

ELIGIBILITY:
Inclusion Criteria:

* Be in good general health based on a physical examination, medical history, vital signs, 12-lead ECG and screening urine and blood tests
* Test negative for recent cannabis use in urine at the screening visit (confirmed by Gas Chromatography (GC)/ Mass Spectrometry (MS) laboratory test) and at clinic admission
* Test negative for other drugs of abuse, including alcohol at the screening visit and at clinic admission
* Demonstrate ability to expectorate 3-5 mL of "native" oral fluid over a 5-minute period
* Not be pregnant or nursing (if female). All females must have a negative serum pregnancy test at the screening visit and a negative urine pregnancy test at clinic admission.
* Have a body mass index (BMI) in the range of 19 to 36 kg/m2
* Blood pressure at Screening Visit does not exceed a systolic blood pressure (SBP) of 150 mmHg or a diastolic blood pressure (DBP) of 90 mmHg
* Have no allergies to any of the ingredients used to prepare cannabis brownies (chocolate, eggs, wheat, etc.).
* Report prior experience inhaling cannabis (either via smoking or vaporization).

Exclusion Criteria:

* History of or current evidence of significant medical or psychiatric illness judged by the investigator to put the participant at greater risk of experiencing an adverse event due to exposure or completion of other study procedures.
* Use of an Over-the-Counter (OTC), systemic or topical drug(s), herbal supplement(s), or vitamin(s) within 14 days of experimental sessions; which, in the opinion of the investigator or sponsor, will interfere with the study result or the safety of the subject.
* Use of a prescription medication (with the exception of birth control prescriptions) within 14 days of experimental sessions; which, in the opinion of the investigator or sponsor, will interfere with the study result or the safety of the subject.
* Use of hemp seeds or hemp oil in any form in the past 3 months.
* Use of dronabinol (Marinol) within the past 6 months.
* History of xerostomia (dry mouth), or the presence of mucositis, gum infection or bleeding, or other significant oral cavity disease or disorder that in the investigator's opinion may affect the collection of oral fluid samples.
* History of clinically significant cardiac arrhythmias or vasospastic disease (e.g., Prinzmetal's angina).
* Abnormal EKG result that in the investigator's opinion is clinically significant.
* Epilepsy or a history of seizures.
* Enrolled in another clinical trial or have received any drug as part of a research study within 30 days prior to dosing

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 23 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2019-06-11 (Actual); Study Completion 2020-02-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ryan Vandrey, PhD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins University School of Medicine, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This was a within-subjects design, so all participants were exposed to all six conditions in a randomized order.
Groups:
- Oral Cannabis 0mg, 10mg, 25mg; Vaporized Cannabis 0mg, 5mg, 20mg: Participants ingested and vaporized THC in the above order in a within-subject crossover design
Period: Overall Study
Arm/Group | Oral Cannabis 0mg, 10mg, 25mg; Vaporized Cannabis 0mg, 5mg, 20mg
Started | 23
Oral 0mg | 22
Oral 10mg | 22
Oral 25mg | 21
Vape 0mg | 20
Vape 5mg | 21
Vape 20mg | 21
Completed | 20
Not Completed | 3

BASELINE CHARACTERISTICS:
Groups:
- All Evaluable Study Completers: Participants received oral (0, 10, 25mg) and vaporized (0mg, 5, 20mg) THC in a randomized within-subject crossover design
Arm/Group | All Evaluable Study Completers
Number analyzed (Participants) | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 28.5 (6.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 17
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 7
  White | 9
  More than one race | 0
  Unknown or Not Reported | 3
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 20

OUTCOME MEASURES:

1. Primary Outcome: Tetrahydrocannabinol (THC) Concentration in Blood
Description: Quantitation of active drug (THC) in whole blood (ng/ml).
Time Frame: 8 hours
Population: This was a within-subjects design, so all participants were exposed to all six conditions in a randomized order.
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Placebo Oral Cannabis | Low-Dose Oral Cannabis | High-Dose Oral Cannabis | Placebo Vaporized Cannabis | Low-Dose Vaporized Cannabis | High-Dose Vaporized Cannabis
Number analyzed (Participants) | 20 | 20 | 20 | 20 | 20 | 20
ng/ml | 0 (0) | 1.78 (1.93) | 3.06 (2.41) | 0 (0) | 9.19 (10.43) | 37.24 (22.36)

2. Secondary Outcome: 11-hydroxy-tetrahydrocannabinol (11-OH-THC)
Description: Quantitation of THC metabolite in blood (ng/ml)
Time Frame: 8 hours
Population: This was a within-subjects design, so all participants were exposed to all six conditions in a randomized order.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Placebo Oral Cannabis | Low-Dose Oral Cannabis | High-Dose Oral Cannabis | Placebo Vaporized Cannabis | Low-Dose Vaporized Cannabis | High-Dose Vaporized Cannabis
Number analyzed (Participants) | 20 | 20 | 20 | 20 | 20 | 20
ng/mL | 0 (0) | 1.7 (1.7) | 2.5 (1.0) | 0 (0) | 0.72 (1.1) | 1.3 (1.1)

3. Secondary Outcome: Tetrahydrocannabinolic Acid (THCCOOH)
Description: Quantitation of THC metabolite in blood (ng/ml).
Time Frame: 8 hours
Population: This was a within-subjects design, so all participants were exposed to all six conditions in a randomized order.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Placebo Oral Cannabis | Low-Dose Oral Cannabis | High-Dose Oral Cannabis | Placebo Vaporized Cannabis | Low-Dose Vaporized Cannabis | High-Dose Vaporized Cannabis
Number analyzed (Participants) | 20 | 20 | 20 | 20 | 20 | 20
ng/mL | 0 (0) | 7.7 (4.5) | 18.4 (9.3) | 0 (0) | 2.2 (2.5) | 5.6 (3.3)

4. Secondary Outcome: Change in Heart Rate
Description: Peak change from baseline
Time Frame: Baseline, 1, 2, 3, 4, 5, 6, 7, and 8 hours post drug exposure
Population: This was a within-subjects design, so all participants were exposed to all six conditions in a randomized order.
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | Placebo Oral Cannabis | Low-Dose Oral Cannabis | High-Dose Oral Cannabis | Placebo Vaporized Cannabis | Low-Dose Vaporized Cannabis | High-Dose Vaporized Cannabis
Number analyzed (Participants) | 20 | 20 | 20 | 20 | 20 | 20
Beats per minute | -0.7 (14.9) | 3.7 (14.8) | 12.2 (14.1) | -1.8 (11.8) | 8.7 (16.9) | 20.8 (21.4)

5. Secondary Outcome: Mean (SD) Peak Change-from-baseline Drug Effect Rating
Description: Subjective rating of drug effect (0-100) at peak effect: between 2 and 5 hours for oral dosing conditions and 0 and 2 hours for vaporized conditions. Higher numbers mean stronger drug effects, where 0 means no drug effect and 100 means extremely strong drug effect.
Time Frame: Up to 5 hours
Population: This was a within-subjects design, so all participants were exposed to all six conditions in a randomized order.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Placebo Oral Cannabis | Low-Dose Oral Cannabis | High-Dose Oral Cannabis | Placebo Vaporized Cannabis | Low-Dose Vaporized Cannabis | High-Dose Vaporized Cannabis
Number analyzed (Participants) | 20 | 20 | 20 | 20 | 20 | 20
Score on a scale | 4.5 (12.5) | 36.9 (31.8) | 59.5 (36.6) | 5.6 (15.4) | 58.2 (37.0) | 84.1 (26.2)

6. Secondary Outcome: Change From Baseline Behavioral Task Performance as Assessed by the DRUID App Score
Description: Composite Global Impairment Score on the DRUID (DRiving Under the Influence of Drugs) App, a measure of behavioral task performance (range 0-100) where lower scores indicate better performance. ≥13-point change (from baseline) on DRUID global impairment score = "impaired"; <13-point change (from baseline) = "not impaired".
Time Frame: 8 hours
Population: This was a within-subjects design, so all participants were exposed to all six conditions in a randomized order.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo Oral Cannabis | Low-Dose Oral Cannabis | High-Dose Oral Cannabis | Placebo Vaporized Cannabis | Low-Dose Vaporized Cannabis | High-Dose Vaporized Cannabis
Number analyzed (Participants) | 20 | 20 | 20 | 20 | 20 | 20
score on a scale | -0.1 (6.5) | 4.5 (9.3) | 12.9 (8.2) | 1.3 (6.9) | 4.7 (8.9) | 10.5 (15.2)

7. Secondary Outcome: Peak Change in Blood Pressure
Description: Systolic and Diastolic blood pressure will be measured at baseline and repeatedly for 8 hours after drug exposure. Outcome is the peak change from baseline assessed within the 8 hour period of assessment.
Time Frame: 8 hours post drug exposure
Population: This was a within-subjects design, so all participants were exposed to all six conditions in a randomized order.
Measure: Mean (Standard Deviation); unit: mm/Hg
Arm/Group | Placebo Oral Cannabis | Low-Dose Oral Cannabis | High-Dose Oral Cannabis | Placebo Vaporized Cannabis | Low-Dose Vaporized Cannabis | High-Dose Vaporized Cannabis
Number analyzed (Participants) | 20 | 20 | 20 | 20 | 20 | 20
mm/Hg
  Systolic BP | 1.1 (13.8) | 1.0 (16.1) | 0.5 (15.4) | -2.4 (13.5) | -2.8 (15.3) | -4.8 (15.6)
  Diastolic BP | -2.3 (11.7) | -0.9 (14.4) | -1.1 (15.2) | 2.8 (12.7) | 2.9 (11.2) | 0.2 (14.0)

ADVERSE EVENTS:
Time Frame: 1 year, 1 month
Description: This was a within-subjects cross-over design. All participants were exposed to all six dose conditions. Exposure was clustered by route of administration (oral vs vaporized) and doses within each route were administered in a randomized order.
Arm/Group | Placebo Oral Cannabis | Low-Dose Oral Cannabis | High-Dose Oral Cannabis | Placebo Vaporized Cannabis | Low-Dose Vaporized Cannabis | High-Dose Vaporized Cannabis
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20 | 0/20 | 0/20 | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20 | 0/20 | 0/20 | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 0/20 | 0/20 | 0/20 | 0/20 | 0/20 | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-05-18): https://cdn.clinicaltrials.gov/large-docs/91/NCT03122691/Prot_SAP_000.pdf
  • Informed Consent Form (2018-06-05): https://cdn.clinicaltrials.gov/large-docs/91/NCT03122691/ICF_001.pdf